CLINICAL TRIAL: NCT01573494
Title: Study of Circulating Tumor Cells Before and After Treatment in Patients With Metastatic Melanoma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-AOI-04
Record Dates: First submitted 2012-03-23; First posted 2012-04-09 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Melanoma
Keywords: Cancer; Melanoma; Circulating Tumor Cells
MeSH Terms: conditions — Melanoma; Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metastatic melanoma patients (Experimental): Sampling of blood before and after chemotherapy
  Interventions: Other: Sampling of blood

INTERVENTIONS:
Other: Sampling of blood — 7,5 ml of blood

SUMMARY:
Circulating tumor cells (CTC) are the subject of increasing interest in clinical oncology as a prognostic factor and predictor of therapeutic response. The detection of CTC by immunomagnetic method has proved its reliability and its usefulness for monitoring breast cancer, colon and prostate in the metastatic and immunomagnetic detection system (CellSearch, Veridex LLC) was approved by the FDA in these indications. However, to date there is no reliable method to detect CTCs in melanoma (CMC). Studies based on PCR amplification of mRNA by reverse specific melanoma is disappointing. Recently, a new detection system of CMC immunomagnetic was presented (CellSearch, Veridex LLC, United States). This system has the advantage of combining immunomagnetic selection step and a step of identifying by immunofluorescence. A preclinical study on serial dilutions of melanoma cells has shown encouraging results. The investigators propose a prospective study of the CellSearch system in patients with melanoma.

Primary objective: To determine the effect of treatment on the number of circulating melanoma cells in patients with metastatic melanoma.

Secondary objectives:

* determine the percentage of patients with metastatic melanoma with melanoma cells circulating
* seek a relationship between the number of circulating melanoma cells and prognosis in patients with metastatic melanoma
* seek a relationship between the change in the number of circulating melanoma cells before / after treatment and tumor response in patients with metastatic melanoma

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 18 years
* Patients with advanced melanoma stage IIIC (unresectable) or stage IV
* Patient not treated or not responding to chemotherapy with chemotherapy session last> 1 month
* Patients who signed informed consent
* Patients presenting no socio-economic, psychological, familial or geographical allow proper understanding of the information leaflet of the protocol or the regular monitoring in the department of dermatology
* Patients with a life expectancy greater than 3 months
* Patients with melanoma measurable by RECIST version 1.1
* Patients with venous good for venipuncture

Exclusion Criteria:

* Patients with contraindication for treatment with chemotherapy or V600E BRAF inhibitor or ipilimumab or have conditions concomitant heavy may interfere with the treatment of metastatic melanoma
* Pregnant women or nursing
* People vulnerable detainees, adults under guardianship or curatorship, minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Measuring the number of circulating melanoma cells/ml in blood | baseline and 3 months
  Measuring the number of circulating melanoma cells/ml in the peripheral blood by the test before and after treatment CellSearch.

SECONDARY OUTCOMES:
number of patients who test positive detection of circulating melanoma cells measured in peripheral blood with the CellSearch test | 3 months
  Calculating the number of patients who test positive detection of circulating melanoma cells measured in peripheral blood with the CellSearch test before and after treatment.
Difference in survival | baseline and 6 months
  Difference in survival between patients depending on the number of circulating melanoma cells/ml before treatment, according to Kaplan-Meier method.
Difference in tumor response | 6 months
  Difference in tumor response between patients according to the variation of circulating melanoma cells/ml before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Damien GIACCHERO, PH, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France